CLINICAL TRIAL: NCT03727256
Title: Recep Tayyip Erdogan University Medical School
Brief Title: Neuromuscular Electrical Stimulation and Ultrasound Therapies , Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gul Devrimsel, Principal Investigator, Recep Tayyip Erdogan University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No sponsor
Record Dates: First submitted 2018-10-22; First posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; neuromuscular electrical stimulation; ultrasound therapy
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 patients (Active Comparator): Patients have grade 2 or 3 knee osteoarthritis ultrasound therapy
  Interventions: Other: ultrasound therapy
- Group 2 patients (Active Comparator): Patients have grade 2 or 3 knee osteoarthritis neuromuscular electrical stimulation application
  Interventions: Other: neuromuscular electrical stimulation application

INTERVENTIONS:
Other: ultrasound therapy — Group 1, ultrasound therapy ;1 watt/cm² dose, 1 MHz, 5 minutes
  Arms: Group 1 patients
Other: neuromuscular electrical stimulation application — Group 2, neuromuscular electrical stimulation application;20 mins/session
  Arms: Group 2 patients

SUMMARY:
To determine the effects of ultrasound therapy and neuromuscular electrical stimulation on the muscle architecture and functional capacity of patients with knee osteoarthritis.

DETAILED DESCRIPTION:
All participants who were satisfied with the inclusion criteria were randomly assigned to one of two study groups: Group 1- ultrasound therapy group; Group 2 - the neuromuscular electrical stimulation group. Group allocation was randomized in two blocks of 30 sealed envelopes without external marks, which were mixed and numbered from 1 to 30, containing a piece of paper with the group allocation. The researchers responsible for outcome measures and ultrasonograhic measurements were blinded to the patients' diagnosis or intervention.

ELIGIBILITY:
1. Inclusion Criteria:

   Clinical diagnosis of knee osteoarthritis
2. Exclusion Criteria:

Cardiovascular diseases

Inflammatory diseases

Infectious diseases

Lower extremity weakness

Tumoral diseases

Knee surgery in the past six months

Intra-articular injection in the past six months

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | 3 weeks
  Pain was assessed using a 0 to 10 visual analogue pain scale, with 0 meaning 'no pain' and 10 meaning 'excruciating pain'.
Western Ontario and McMaster Universities Arthritis Index | 3 weeks
  The WOMAC (Westren Ontario and McMaster Universities) index is used to assess patients with osteoarthritis of the hip or knee using 24 parameters.To assess pain, stiffness, and physical function in patients with hip and / or knee osteoarthritis, Minimum total score: 0, maximum total score: 96.Disability scores increase as Womac osteoarthritis index scores increase.
15 meter walking test | 3 weeks
  The patients were asked to walk as fast as possible along a level, unobstructed corridor on the command "go." The patients stood before the starting line. A hand-held stopwatch was started as the subjects passed a predetermined start mark and stopped as they passed a second mark 15meter from the start mark.Walking duration was determined as second before and after treatment
Muscle measurements were made before and after treatment. | 3 weeks
  Ultrasonography was used to measure muscle thickness, pennation angle and fascicle length. Muscle thickness was measured as the mean distance between the superficial and deep aponeurosis at both image muscles. The distance between the intersection composed of the superficial aponeurosis and muscle fascicle, and the intersection composed of the deep aponeurosis and muscle fascicle was defined as muscle fascicle length. The results was measured as millimeter.The angle between the muscle fascicle and deep aponeurosis was defined as Pennation angle.

CONTACTS AND LOCATIONS:
Overall Officials: GUL DEVRIMSEL, Study Director — Dr.
Locations (1):
- Gul Devrimsel, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No